CLINICAL TRIAL: NCT04777318
Title: Comparison of the Effects of Muscle Energy Technique and Mobilization Techniques on Cervical Proprioception and Motor Control in Patients With Cervical Spondylosis: A Randomized Controlled Study
Brief Title: Comparison of the Effects of Different Manual Therapy Techniques in Patients With Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Buse Sezerel, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0041
Record Dates: First submitted 2021-02-19; First posted 2021-03-02 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Cervical Spondylosis
Keywords: Cervical Spondylosis; Proprioception; Manual Therapies
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Masking Description: Individuals between the ages of 40-65 diagnosed with cervical spondylosis will be included in the study. The sample size was determined as 66 subjects, 22 in each group, under the assumption that the one-way ANOVA test would be applied in the comparison between groups and the effect size would be f = 0.40, α = 0.05, β = 0.20.
  Considering the possibility of using the nonparametric equivalent instead of the parametric ANOVA test in the analyzes that will start after the data collection phase, this initial sample size was increased by 15% and corrected to 76 people. Considering that there may be people who may leave the study, this sample size was increased by 25% and the final sample size was determined as 96 people.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional physiotherapy (Experimental): The individuals in the control group was taken in a total of 12 sessions of conventional physiotherapy program for 4 weeks, 3 days a week.
  Interventions: Other: Conventional physiotherapy
- Muscle Energy Technique (MET) (Experimental): In addition to the conventional physiotherapy program of 12 sessions for 4 weeks, 3 days a week, muscle energy technique was applied to the individuals in the second group.
  Interventions: Other: Conventional physiotherapy and Muscle Energy Technique
- Cervical Mobilization Techniques (CMT) (Experimental): In the third group, cervical mobilization techniques was applied in addition to the conventional physiotherapy program for a total of 12 sessions for 4 weeks, 3 days a month.
  Interventions: Other: Conventional physiotherapy and Cervical Mobilization Techniques

INTERVENTIONS:
Other: Conventional physiotherapy — A total of 12 sessions of conventional physiotherapy program for 4 weeks were applied 3 days a week. The conventional physiotherapy program included 20 min hotpack , 10 min ultrasound, 20 min conventional (Transcutaneous electrical nerve stimulation) TENS application.
  Arms: Conventional physiotherapy
Other: Conventional physiotherapy and Muscle Energy Technique — In addition to conventional therapy, the muscle energy technique was applied to the individuals in the second group at the same frequency. Muscle energy technique was applied to the upper trapezius, sternocleidomastoideus , scalene (anterior-medius-posterior) and levator scapula muscles. According to the MET post-isometric relaxation method, each muscle was applied as one set (each set includes three repetitions). The patient was asked to perform a 7-second isometric contraction corresponding to 20% of the maximum isometric contraction force in the area where the restriction was felt. After the application, the patient was asked to breathe and relax, and the neck was brought back to the barrier point and the technique was repeated.
  Arms: Muscle Energy Technique (MET)
Other: Conventional physiotherapy and Cervical Mobilization Techniques — Cervical mobilization techniques were also applied to the individuals in the third group in addition to conventional physiotherapy at the same frequency. In the first few sessions, bridging and manual traction techniques were applied in 3-5 repetitions. In the next sessions, in addition to these techniques, rotation with 3-5 repetitions of manual traction, anteroposterior sliding with traction and cervical lateral shift techniques were applied. Vertebrobasilar InsufficiencyTest was applied to all participants to determine the appropriateness of cervical mobilization. Before mobilization, a deep friction massage was applied on painful spasmic nuchal muscles for 3-4 minutes in order to increase blood circulation and relax tense tissues.
  Arms: Cervical Mobilization Techniques (CMT)

SUMMARY:
Proprioceptive sensitivity decreases in individuals with neck pain compared to those without neck pain. While organizing the treatment program of patients with neck pain, evaluation of cervical proprioception and its addition to the treatment have gained importance.

The aim of the study was to examine the effects of muscle energy technique applied to patients with chronic neck pain on cervical proprioception and motor control and to compare the results of muscle energy technique application with cervical mobilization techniques.

DETAILED DESCRIPTION:
Cervical spondylosis (SS) is defined as chronic disc degeneration due to aging caused by degenerative changes in the muscles, tendons, joints or bones of the neck or shoulder.

The etiology of cervical spondylosis includes various factors such as bad posture, anxiety, depression, neck strain, and overload in sports or occupational activities. Proprioception is defined as sensory feedback that contributes to muscle sensation, postural balance and joint stability. It is possible that loss of cervical proprioception and motor control affect segmental stability. This increases the risk of injury following minor trauma. It has been reported that proprioceptive sensitivity is worse in individuals with neck pain compared to those without neck pain, and the degree of the disorder is related to the severity of pain. Some evidence-based studies have shown that manual techniques improve proprioception and motor control.

It has been shown that Muscle Energy Technique (MET), which has gained popularity in recent years, increases cervical joint mobility and reduces pain in patients with chronic neck pain. MET is a form a manual therapy which uses a muscle's own energy in the form of gentle isometric contractions to relax the muscles via autogenic or reciprocal inhibition mechanism. It has been reported that MET stimulates joint proprioceptors, creates a different movement activity in the area of proprioceptive disorder and allows the central nervous system to normalize proprioceptive and motor coordination in this segment. The effect of MET on cervical proprioception in patients with cervical spondylosis has not been investigated yet.

Active participation of the patient in movement is extremely important in proprioceptive feedback, motor control and motor learning. For this reason, it is thought that investigating the effect of MET, which includes active muscle contractions of the patient, on proprioceptive sense and comparing the results with passive applications (manipulation or mobilization) will be useful in determining the optimal treatment method in cervical spondylosis.

ELIGIBILITY:
Inclusion Criteria:

* Presence of neck pain of Visual Analog Pain Scale (VAS) ≥ 2 in at least one direction lasting more than three months
* Not having received conservative treatment in the last 6 months

Exclusion criteria

* Pain or numbness that spreads to the arms
* Having a cervical region surgery
* Having musculoskeletal problems such as shoulder impingement or thoracic outlet syndrome
* Having a contraindication to cervical mobilization (VBI, myelopathy, inflammatory arthropathy, malignancy, etc.)
* Using analgesic drugs
* People who cannot adapt to study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Neutral head position test (NBPT) | 4 week
  NBPT as assessed using the CROM (cervical range of motion) device, which is a special goniometer for the neck. NBPT was started when the cervical region is in a neutral position, the individual was asked to turn his head completely to the left or right and return to the neutral position in a controlled manner. The angular difference was recorded in degrees.
Target head position test (HBPT) | 4 week
  CROM device was used for HBPT evaluation. The researcher passively moved the person's head to the pre-determined target position, 50% of the maximum range of motion. The head was held in the target position for 3 seconds (sec), then the person was asked to move the head to the neutral position first and then actively move it back to the target position. The angular difference was recorded in degrees.
Cervical region movement sensation | 4 week
  The laser pointer was fixed on the individual's head. The person sat on a chair 1 m away from the ZZ pattern, which was transferred to a 13 cm high A4 paper with 23.4 horizontal and 26.6 long diagonal stripes fixed to the wall.
  The pattern has five thin additional lines every 5 mm from the baseline to differentiate the five deviation zones. The test was recorded with a camera 50 cm from the center of the pattern. Individuals will be asked to follow the bands of the pattern as accurately and as quickly as possible, starting from the center of the pattern, and the test was considered complete when it returns to its starting position. After the test, video files were examined at 1/8 of the normal speed, to be used in analysis; time, error frequency and error size were calculated.
Neck pain intensity | 4 week
  Visual analog scale (VAS) was used to neck pain intensity during resting and activity.

SECONDARY OUTCOMES:
Craniocervical Flexion Test (CCFT) | 4 week
  CCFT is used to evaluate the activation and static endurance of the deep flexor muscles of the cervical region. CCFT is also defined as the motor control test of the cervical region. The test was performed using Stabilizer Pressure Biofeedback (Chattanooga Stabilizer). The patient was positioned in the supine position, with the cervical region in neutral position and the biofeedback pressure unit was placed in the suboccipital space. The pressure cell was inflated to 20 mmHg in order to support cervical lordosis. Then, the individual was instructed to perform a posterior tilt movement by increasing the pressure at 5 different levels (22, 24, 26, 28 and 30 mmHg.), by following the monitor of the device. After teaching the movement, the person was asked to perform 10 contractions lasting 10 seconds at each level. The person moved the next level after each successful attempt and was given a 10-second rest period between repetitions.
Cervical flexor muscle endurance | 4 week
  Cervical flexor muscle endurance was evaluated with the patient lying in the supine position with the knees flexed. The person was asked to press their chin back and lift their head approximately 2.5 cm from the bed while maintaining this position. The time the individual maintained the position was recorded in seconds.
Cervical extensor muscle endurance | 4 week
  The cervical extensor muscle endurance was evaluated with the patient lying face down and the head hanging from the bed. A belt was passed over the ears of the individuals and weight was tied at the end. The weight was been 2.32 kg for women and 4 kg for men. The individual was asked to bring his head to a neutral position and to maintained this position. The time the individual maintained the position was recorded in seconds.
Dynamic balance | 4 week
  It was evaluated using the Y balance test. The reach distance in the anterior, posteromedial and posterolateral transport directions were recorded. People was asked to reach the furthest point with the other foot while trying to maintain balance with the dominant foot on the wooden platform while the hands are on the waist. 3 repetitions of reaching out in 3 directions were recorded. Mixed reach distance; was calculated using the formula [(maximum anterior + maximum posteromedial + maximum posterolateral) / (3 x lower extremity length)] x 100.
Static balance | 4 week
  It was evaluated with both eyes closed and eyes open using the single leg balance test (SLBT). Individuals was asked to cross their arms at chest level and focus on a point on the wall. The test started when the foot was lifted off the ground and the time it remained in this position was recorded in seconds using a stopwatch.
Neck pain related disability | 4 week
  The Copenhagen Neck Functional Scale (KBFSÖ) is a scale evaluating the effect of neck pain related disability. It has excellent internal consistency and test-retest reliability and good validity with pain scale. The scale consists of 15 items. The total score of the questionnaire can range from 0 (no neck pain effect) to 30 (worst possible effect). Items 1 and 5 directly assess pain intensity; Items 2, 3, 4, 5, 7, 8, 9, and 10 assess disability during daily activities; and Articles 6, 9, 11, 13 and 14 focus on social interactions and recreational activities. The last item 15 evaluates the patient's perception of the future impact of neck pain. The questions were answered individually as yes (0 points), sometimes (1 point) and no (2 points). The total score was recorded for use in analysis.

CONTACTS AND LOCATIONS:
Overall Officials: İNCİ YÜKSEL, Prof. Dr., Study Director — Eastern Mediterranean University
Locations (1):
- Buse Sezerel, Famagusta, Cyprus